CLINICAL TRIAL: NCT01092390
Title: "Go Fish"Omega-3 Fatty Acid Supplementation in Diabetic Kidney Disease
Brief Title: Go Fish: Omega-3 Fatty Acid Supplementation in Diabetes-Related Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Edgar R. Miller, III, PI, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21DK080372 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes
Keywords: randomized trial; omega three fatty acids
MeSH Terms: conditions — Diabetes Mellitus | interventions — Omacor; Fish Oils; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lovaza (Experimental): 4 grams per day
  Interventions: Dietary Supplement: Lovaza (fish oil)

INTERVENTIONS:
Dietary Supplement: Lovaza (fish oil) — 4 grams per day
  Other Names: fish oil (generic); omega three fattay acids (generic)

SUMMARY:
In this application the investigators describe plans for a randomized controlled cross-over trial to determine the effects of omega-3 fatty acid supplementation on urine protein excretion in 30 adults with diabetes (NIDDM) and kidney disease defined by the presence of proteinuria.

DETAILED DESCRIPTION:
Diabetes is the most common cause of end-stage kidney disease in the United States. Half of patients with diabetes develop kidney disease. The benefits of omega-3 fatty acids have been shown in animal models of kidney injury. Mechanistic studies of omega-3 fatty acid supplements support biological plausibility: omega-3 supplements have been shown to improve vascular reactivity, lower oxidative stress, reduce inflammation, and have beneficial effects on the metabolism of eicosanoids favoring synthesis of vasodilatory prostaglandins and thromboxanes. However, in spite of overwhelming evidence for a potential benefit of dietary omega-3 fatty acids at preventing or slowing progression of kidney disease for adults with NIDDM, clinical trials providing evidence to support recommendations of supplementation are lacking.

The current recommendation for omega-3 intake for adults, one gram/day of DHA+EPA, is based on evidence for cardiovascular disease risk (CVD) reduction. Whether omega-3 fatty acid prevents or slows progression of diabetic kidney disease, whether the current recommended dose is adequate to modify disease, or whether a higher dose should be recommended, needs to be determined.

In this setting, we propose to conduct a randomized placebo-controlled cross-over clinical trial to determine the effects of a daily dose of omega-3 fatty acid supplementation (4.0 g/day) compared with placebo on urine protein excretion and biomarkers of kidney injury and function in adults with diabetes and proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Participants have a diagnosis of diabetes (either oral medication or diet controlled)
* Have an average systolic blood pressure (SBP) <150 and diastolic blood pressure (DBP) <90 mmHg
* Have quantified proteinuria -- urine albumin/creatinine ratio of > 17 mg/g (men) and >25 mg/g (women) (i.e. at least microalbuminuria).
* Participants must be on stable doses of antihypertensive, hypoglycemic, and lipid lowering medications for a minimum of two months prior to randomization. Participants must agree to stay on stable doses of diabetes, antihypertensive and lipid medication for the duration of the study.

Exclusion Criteria:

* Major exclusion criteria will be poorly controlled diabetes (Hemoglobin A1c >9%)
* Use of insulin
* Use of fish oil supplements or are unwilling to stop fish oil supplements one month prior to randomization and refrain from the supplements during the study
* Stage 4 or stage 5 CKD or a screening urine protein/creatinine ratio of >2.5.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
urine protein excretion | end of 2 six week periods (crossover)
  Primary Specific Aim To determine the effects of omega-3 fatty acid supplementation on urine protein excretion and surrogate markers of kidney injury including: serum beta-microglobulin and cystatin C (biomarkers of GFR) and urine neutrophil gelatinase-associated lipocain (NGAL a.k.a. lipocalin-2), kidney injury molecule-1 (KIM-1), and interleukin-18 (IL-18) (biomarkers of tubular reabsorption impairment and inflammation).

SECONDARY OUTCOMES:
Biomarkers of oxidation and inflammation | end of 2 six week periods (crossover)
  To determine the effects of omega-3 supplements on markers of oxidations (urine isoprostanes) and inflammation (serum C-reactive protein (hsCRP), RBC fatty acids .

CONTACTS AND LOCATIONS:
Overall Officials: Edgar R Miller, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, 1849 Gwynn Oak Ave, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Miller ER 3rd, Juraschek SP, Anderson CA, Guallar E, Henoch-Ryugo K, Charleston J, Turban S, Bennett MR, Appel LJ. The effects of n-3 long-chain polyunsaturated fatty acid supplementation on biomarkers of kidney injury in adults with diabetes: results of the GO-FISH trial. Diabetes Care. 2013 Jun;36(6):1462-9. doi: 10.2337/dc12-1940. Epub 2012 Dec 28. PMID 23275364